CLINICAL TRIAL: NCT03873571
Title: An Observational Study to Examine the Iron Treatment in Pregnant Women With Anaemia
Brief Title: Adherence of Iron Succinylate Therapy in Pregnancy
Acronym: ARTEMIS
Status: Withdrawn | Type: Observational
Why Stopped: Modification of clinical development plan
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-IRPS-EL-96
Record Dates: First submitted 2019-03-12; First posted 2019-03-13 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Pregnancy Related; Pregnancy Anemia; Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to the World Health Organization (WHO), anemia is the most common disease, affecting >1.5 billion people worldwide. Furthermore, iron deficiency anemia (IDA) accounts for 50% of cases of anemia. IDA is common during pregnancy and the postpartum period, and can lead to serious maternal and fetal complications. Measurement of serum ferritin has the highest sensitivity and specificity for diagnosis of IDA unless there is a concurrent inflammatory condition. The lower threshold value for hemoglobin (Hb) in pregnant women is <11 g/dL during the 1st and 3rd trimesters, and <10.5 g/dL during the 2nd trimester. In postpartum period a Hb concentration <10 g/dL indicates clinically significant anemia. Oral iron therapy is given as the first-line treatment for IDA.

DETAILED DESCRIPTION:
Measurement of serum ferritin has the highest sensitivity and specificity for diagnosis of IDA unless there is a concurrent inflammatory condition. The lower threshold value for hemoglobin (Hb) in pregnant women is <11 g/dL during the 1st and 3rd trimesters, and <10.5 g/dL during the 2nd trimester. In postpartum period a Hb concentration <10 g/dL indicates clinically significant anemia.

Oral iron therapy is given as the first-line treatment for IDA. There are several direct and indirect methods to assess adherence to medications, each method has advantages and limits. Many studies have shown that pill counting is more accurate than self-reported adherence.We will investigate the adherence to iron supplementation in pregnant women by using a self-reported adherence questionnaire named SMAQ (Simplified Medication Adherence Questionnaire)

Simplified Medication Adherence Questionnaire (SMAQ) Knobel H; Juega J; Carmona A; Kindelan JM; Ruiz I; Gonzalez J; Collazos J; Casado JL; Alonso J; Ocampo A SMAQ is used to assess non-adherent patients. The six-item SMAQ has been developed to assess adherence in HIV-infected patients, and may be applied in most clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* Anaemia
* Iron treatment before 3 months of pregnancy
* Informed Consent
* Compliant with study procedures

Exclusion Criteria:

* Iron treatment after 3 months of pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with anaemia treated with iron succinylate
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | 9 months
  SMAQ (Simplified Medication Adherence Questionnaire) rating

CONTACTS AND LOCATIONS:
Locations (1):
- Iaso Hospital, Athens, Greece